CLINICAL TRIAL: NCT04975750
Title: Early Prevention of Sick Leave at the Workplace: Design of a Cluster-randomized Controlled Trial of a Problem-solving Intervention Among Employees With Common Mental Disorders
Brief Title: A Problem Solving Intervention Involving Employees at Risk of Sick Leave Due to Common Mental Disorders
Acronym: PRIME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: AFA Insurance (Industry)
Responsible Party: Principal Investigator, Elisabeth Björk Brämberg, PhD, Docent, Associate Professor, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-3084/2019
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Problem solving intervention (Experimental): Problem solving as developed by Nexu and colleguages. First-line managers are trained in the problem solving intervention (1 1/2 day). Thereafter, they apply the problem-solving in 2 - 5 meetings (about 30 - 45 min each) with employees at risk of future sick leave due to common mental disorders.
  Interventions: Behavioral: Problem solving intervention
- Care as usual (Active Comparator): First-line managers participate in a 3 hour lectur including a brief overview about worker health, occupational stress and the mismatch model and self-efficacy. Thereafter, they provide care-as-usual to employees at risk of future sick leave due to common mental disorders.
  Interventions: Behavioral: Care as usual

INTERVENTIONS:
Behavioral: Problem solving intervention — The intervention focuses on the individual employee and his/her work situation and work-private life balance. The following steps are implemented: inventory and prioritization of problems; brainstorming options and solutions; formulation of an action plan; evaluation, and follow-up. The intervention is carried out in about 3 planned meetings (30 - 45 min) between the manager and the employee. However, given the lack of research regarding the intervention delivered to this specific population and which dose that should be considered as beneficial as well as the complexities of the identified problems, the number of meetings is not specified
  Arms: Problem solving intervention
Behavioral: Care as usual — The managers and the employee have meetings regarding the employee and his/her work situation and work-private life balance. However, the managers are not educated in and do not use the problem solving intervention. They are instead instructed to use their usual procedures.
  Arms: Care as usual

SUMMARY:
The overall aim of this randomized controlled trial is to evaluate the effectiveness of a problem-solving intervention for the prevention of sick leave among employees with early signs of CMDs. The intervention is delivered by first-line managers and a 30% reduction in sick leave days is expected in the experimental condition compared to treatment-as-usual, during the 12- months follow-up.

DETAILED DESCRIPTION:
The overall aim of this randomized controlled trial is to evaluate the effectiveness of a problem-solving intervention for the prevention of sick leave among employees with early signs of CMDs. The intervention is delivered by first-line managers and a 30% reduction in sick leave days is expected in the experimental condition compared to treatment-as-usual, during the 12- months follow-up.

In an alongside process evaluation on the intervention's core activities, i.e. identification of early signs of CMDs, training of first-line managers in problem-solving and communication, we will:

* evaluate whether and to what extent it was possible for the first-line managers to adhere to the intervention's protocol,
* investigate the association between the intervention's core activities and number of sick leave days,
* identify the facilitators and barriers to the intervention among first-line managers and employees and,
* explore the first-line manager's organizational resources supporting their general managerial work.

The study will be conducted in private sector companies, among first-line managers and blue-collar workers. The outcomes will be evaluated on both cluster- and individual participant level.

ELIGIBILITY:
Inclusion Criteria:

* scoring with a cut-off ≥3 points on the GHQ-12, or a positive answer on the question on risk of SA, namely employee believes that he/she will receive a sickness certification due to stress, anxiety, or depression the following 12 months.
* negative answer on the question on bullying, namely employee has not been exposed to bullying by his or her first line manager.
* understand written and spoken Swedish.

Exclusion Criteria:

* Ongoing sick leave (full- or part-time), leave of absence, pregnancy.
* Sick leave ≥14 calendar days during the last 3 months due to CMD.
* At the time for inclusion planned long-term absence during the coming year (for example parental leave, new job, retirement).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sick leave | From baseline until 12 months
  The total number of days on sick leave due to CMDs (including the first 14 calendar days compensated by the employer) during the 12 month follow-up period

SECONDARY OUTCOMES:
Work performance | From baseline until the 12-month follow-up
  Evaluated by two items: one item about impairment of work performance due to health problems (presenteeism), and one item about impairment of work performance due to work environment problems. Karlsson ML, Bergstrom G, Bjorklund C, Hagberg J, Jensen I: Measuring production loss due to health and work environment problems: construct validity and implications. J Occup Environ Med 2013, 55(12):1475-1483.
  Scale ranging from 0 to 10, higher scores indicate worse outcome.
Work ability | From baseline until the 12-month follow-up
  Measured by three items of the Work Ability Index (WAI) Perceived work ability in relation to physcial and mental demands of the work are measured by a five-point scale, ranging from "very bad" to "excellent".
  The employee's beliefs about workability is measured by a three-point sca,e ranging from "unlikely" to "relatively certain".
Self-rated general health | From baseline until the 12-month follow-up
  Measured with a single item from the Short-Form Health Survey, with a five-point response scale, ranging from 1 (excellent) to 5 (bad).
Depressive and anxiety symptoms | From baseline until the 12-month follow-up
  Severity of depressive and anxiety symptoms are assessed by the Hospital Anxiety and Depression Scale.
  The response format is a 4-point scale, ranging from 0 to 3, with higher scores indicating higher levels of depressive or anxiety symptoms.
Self-rated exhaustion | From baseline until the 12-month follow-up
  Assessed by four items of the Self-rated exhaustion disorder (s-ED) scale, with the response format yes/no. Reference: Glise K, Hadzibajramovic E, Jonsdottir IH, Ahlborg G Jr. Self-reported exhaustion: a possible indicator of reduced work ability and increased risk of sickness absence among human service workers. Int Arch Occup Environ Health. 2010 Jun;83(5):511-20. doi: 10.1007/s00420-009-0490-x. Epub 2009 Nov 27. PMID: 19943058.
Psychosocial work environment | From baseline until the 12-month follow-up
  The Copenhagen Psychosocial Questionnaire (COPSOQ) III, Swedish standard version, is used for assessing demands at work (3 questions quantitative and 3 questions emotional demands, responses are given on a five-point scale ranging from Always (100) to Never/hardly ever (0). Higher scores mean a worse outcome); for assessing interpersonal relations and leadership (2 questions recognition and 3 questions quality of leadership, responses are given on a five-point scale from To a very large extent (100) to To a very small extent, Higher scores mean a better outcome), and for assessing work-individual interface (3 questions commitment to the workplace and 3 questions work-life conflict, responses are given on a five-point scale from To a very large extent (100) to To a very small extent, Higher scores mean a better outcome for Commitment to the workplace, while higher scores mean a worse outcome for Work-life conflict).
Work stress | From baseline until the 12-month follow-up
  Single Item stress question (SISQ) with a five-poing response scale ranging from 1 ("not at all") to 5 ("very much"). Arapovic-Johansson B, Wåhlin C, Kwak L, Björklund C, Jensen I: Work-related stress assessed by a text message single-item stress question. Occupational medicine (Oxford, England) 2017, 67(8):601-608.
Life-work conflict | From baseline until the 12-month follow-up
  Impact of private life on work is measured by a single item question from the General Nordic Questionnaire with the response anchors "Very seldom or never" to "very often or always".

OTHER OUTCOMES:
General self-efficacy | From baseline until the 12-month follow-up
  The employee's beliefs in his/her ability to cope with the current situation, mobilize motivation and to act upon demands in different situations, measured by a Swedish validated version of General self-efficacy scale, responses are given on a four-point scale ranging from 1 ("not at all true" to 4 ("exacly true"). Reference: Love J, Moore CD, Hensing G: Validation of the Swedish translation of the General Self-Efficacy scale. Qual Life Res 2012, 21(7):1249-1253.) as well as by a single item measure of general self-efficacy (Williams G, Smith A: Using Single-Item Measures to Examine the Relationships between Work, Personality, and Well-Being in the Workplace. Psychology 2016, 7(6):753-767.
Manager support | From baseline until the 12-month follow-up
  Measured by the two questions of the Social support from supervisor subscale from the The Copenhagen Psychosocial Questionnaire (COPSOQ) III, Swedish standard version. Responses are given on a five-point scale ranging from Always (100) to never/hardly ever (0). Higher scores mean a better outcome.
Job control | From baseline until the 12-month follow-up
  Job control is measured by the four questions of the Influence at work subscale from The Copenhagen Psychosocial Questionnaire (COPSOQ) III, Swedish standard version. Responses are given on a five-point scale ranging from Always (100) to Never/hardly ever (0). Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Björk-Brämberg@ki.se, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Bjork Bramberg E, Arapovic-Johansson B, Bultmann U, Svedberg P, Bergstrom G. Prevention of sick leave at the workplace: design of a cluster-randomized controlled trial of a problem-solving intervention among employees with common mental disorders. BMC Public Health. 2021 Sep 26;21(1):1756. doi: 10.1186/s12889-021-11786-6. PMID 34565357